CLINICAL TRIAL: NCT03130699
Title: Dulce Digital-Me: An Adaptive mHealth Intervention for Underserved Hispanics With Diabetes
Acronym: DD-Me
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: University of California, San Diego (Other); San Diego State University (Other)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corporate Vice President, Scripps Whittier Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK112322-01A1 (NIH)
Record Dates: First submitted 2017-04-24; First posted 2017-04-26 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; mHealth; Medical Assistant; Automated; Adaptive Feedback; Self-Management Support; Hispanics; HbA1c; Cyberinfrastructure; Federally-Qualified Health Centers; Cost-Effectiveness; T2DM; Pay-for-Performance; Medication Adherence; LDL-C; Systolic Blood Pressure; Text Messaging
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dulce Digital (Experimental): The first of the three arms of the parallel design: The group of participants randomly assigned to this arm of the study receives one-size-fits-all educational text messages, with patient monitoring and transmission of blood glucose values.
  Interventions: Behavioral: Dulce Digital
- Dulce Digital-Me (Automated Delivery) (Experimental): The second of the three arms of the parallel design: The group of participants randomly assigned to this arm of the study receives educational text messages, with patient monitoring and transmission of blood glucose values, plus personalized goal-setting and tailored feedback delivered via automated algorithm-driven messaging, incorporated into existing primary care team processes.
  Interventions: Behavioral: Dulce Digital-Me (Automated Delivery)
- Dulce Digital-Me (Medical Assistant) (Experimental): The third of the three arms of the parallel design: The group of participants randomly assigned to this arm of the study receives educational text messages, with patient monitoring and transmission of blood glucose values, plus personalized goal-setting and tailored feedback delivered by Medical Assistants, incorporated into existing primary care team processes.
  Interventions: Behavioral: Dulce Digital-Me (Medical Assistant)

INTERVENTIONS:
Behavioral: Dulce Digital — One-size-fits-all educational text messages, with patient monitoring and transmission of blood glucose values.
  Arms: Dulce Digital
Behavioral: Dulce Digital-Me (Automated Delivery) — Educational text messages, with patient monitoring and transmission of blood glucose values, plus personalized goal-setting and tailored feedback delivered via automated algorithm-driven messaging, incorporated into existing primary care team processes.
  Arms: Dulce Digital-Me (Automated Delivery)
Behavioral: Dulce Digital-Me (Medical Assistant) — Educational text messages, with patient monitoring and transmission of blood glucose values, plus personalized goal-setting and tailored feedback delivered by Medical Assistants, incorporated into existing primary care team processes.
  Arms: Dulce Digital-Me (Medical Assistant)

SUMMARY:
This study will compare Dulce Digital (i.e., the investigators' proven-effective combination of "one-size-fits-all" educational text messages and nurse monitoring of patient-transmitted blood glucose values) and Dulce Digital-Me (DD-Me), an adaptive/dynamic mHealth (mobile health) intervention that is tailored to individuals' needs and behavioral progress, in improving diabetes clinical control, adherence, and patient-provider communication in Hispanics - an at-risk, understudied population that experiences disparities in diabetes prevalence and outcomes. These striking disparities in the growing and aging US Hispanic population have taxed the US healthcare system, while significantly reducing quantity and quality of life for millions of individuals. By offering an innovative, scalable, and sustainable approach that seamlessly integrates several mHealth technologies into existing primary care team processes to improve the health of Hispanics (and eventually, other at-risk, underserved groups), DD-Me has strong potential to significantly impact public health.

DETAILED DESCRIPTION:
Individuals of low socioeconomic (SES) and ethnic minority status, including Hispanics, the largest U.S. ethnic minority group, are disproportionately affected by diabetes. Poor healthcare access and cultural barriers prevent optimal care, adherence, and clinical benefit, thus placing Hispanics at high risk for costly diabetes complications. The investigators' established academic-healthcare-community partnership has unique experience in developing and testing innovative, cost-effective, and sustainable chronic care interventions to reduce disparities and improve health in underserved communities. The investigators recently developed Dulce Digital (i.e., "one-size-fits-all" educational text messages, with nurse monitoring of patient-transmitted blood glucose values), which improved glycemic control across 6 months, relative to usual care in a recent randomized controlled trial (RCT) of N=126 Hispanic patients with poorly controlled type 2 diabetes (T2DM). The process evaluation for this trial indicated that Dulce Digital was both feasible and acceptable from patient and provider perspectives; however, patients expressed a preference for a more individualized intervention, and providers requested an even greater focus on health behavior change. Thus, the proposed RCT will examine the comparative effectiveness of Dulce Digital versus "Dulce Digital-Me" (DD-Me) in N=414 Hispanic adults of low SES with poorly controlled T2DM from Neighborhood Healthcare, a San Diego Federally-Qualified Health Center. Guided by patient and provider feedback, DD-Me includes Dulce Digital components plus personalized goal-setting and feedback that is responsive to the individual's needs and preferences. The DD-Me adaptive feedback component will be informed by the Resources and Support for Self-Management Model and Operant Conditioning Theory, and based on the individual's progress on intermediate behavioral targets (i.e., medication adherence assessed by wireless sensor; brief mobile phone-based assessments of diet, physical activity, stress). Feedback will be delivered via algorithm-driven automated messaging in 50% of DD-Me participants and by the care team medical assistant in the remaining half to determine the feasibility and acceptability (given the purported cultural relevance of interpersonal relationships in the Hispanic culture), and the comparative effectiveness and cost of each delivery method. Changes in indicators of diabetes clinical control [i.e., glycosylated hemoglobin (HbA1c) low density lipoprotein cholesterol (LDL-C), systolic blood pressure (SBP)], patient-provider communication, and patient adherence (i.e., to medication and other diabetes self-management behaviors) will be evaluated across twelve months. Thorough process and cost-effectiveness analyses will evaluate the scalability and sustainability potential of DD-Me. This comparative evaluation of two mHealth approaches will elucidate how technology can be integrated most effectively and efficiently within existing nurse-led chronic care approaches to meet the complex needs of underserved individuals with poorly controlled T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified Hispanic/Latino
2. 18 years or older
3. Registered patient of a Neighborhood Healthcare Clinic
4. Diagnosed with T2DM (Type 2 Diabetes Mellitus)
5. HbA1c ≥ 8.0% and/or SBP ≥ 160 mmHg, and/or LDL-C ≥ 100 mg/dL in the last 30 days

Exclusion Criteria:

1. Severe illness precluding regular clinic visits
2. Pregnant or lactating
3. Type 1 or gestational diabetes
4. Lack of minimal literacy
5. Plans to relocate
6. Severe auditory or visual problems
7. Primary language other than Spanish or English
8. Unwilling to carry a mobile phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2021-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute; Linda Gallo, PhD, Principal Investigator — San Diego State University
Locations (2):
- United States (2):
  - Scripps Mercy Chula Vista, Chula Vista, California
  - Scripps Whittier Diabetes Institute, La Jolla, California

REFERENCES:
- [Derived] Philis-Tsimikas A, Fortmann AL, Clark T, Spierling Bagsic SR, Farcas E, Roesch SC, Schultz J, Gilmer TP, Godino JG, Savin KL, Chichmarenko M, Jones JA, Sandoval H, Gallo LC. Dulce Digital-Me: results of a randomized comparative trial of static versus adaptive digital interventions for Latine adults with diabetes. Ann Behav Med. 2025 Jan 4;59(1):kaae077. doi: 10.1093/abm/kaae077. PMID 39707158
- [Derived] Philis-Tsimikas A, Fortmann AL, Godino JG, Schultz J, Roesch SC, Gilmer TP, Farcas E, Sandoval H, Savin KL, Clark T, Chichmarenko M, Jones JA, Gallo LC. Dulce Digital-Me: protocol for a randomized controlled trial of an adaptive mHealth intervention for underserved Hispanics with diabetes. Trials. 2022 Jan 28;23(1):80. doi: 10.1186/s13063-021-05899-x. PMID 35090520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2017 and March 2020, the study enrolled 310 Hispanic adults with low income and poorly managed type 2 diabetes from a San Diego County Federally Qualified Health Center.
Pre-assignment Details: The target sample size based on power analysis was N=414. Enrollment started October 31, 2017 was paused on March 13, 2020, and then concluded early due to the COVID-19 pandemic. Because the design accommodated at 30% attrition rate, sample size was adequate for analysis of outcomes.
Period: Overall Study
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistant)
Started | 107 | 106 | 97
Completed | 67 | 66 | 65
Not Completed | 40 | 40 | 32
Not completed — Lost to Follow-up | 34 | 37 | 26
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Withdrawal by PI | 1 | 2 | 5
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Hispanic adults with low income and poorly managed type 2 diabetes are enrolled from a San Diego County Federally Qualified Health Center.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistant) | Total
Number analyzed (Participants) | 107 | 106 | 97 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.22 (10.7) | 53.21 (10.26) | 51.90 (9.49) | 52.11 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 73 | 67 | 216
  Male | 31 | 33 | 30 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 107 | 106 | 97 | 310
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 0 | 4
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 2 | 1 | 0 | 3
  White | 42 | 37 | 27 | 106
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 56 | 64 | 68 | 188
Region of Enrollment [Number; unit: participants]
  United States | 107 | 106 | 97 | 310
Less than High School Education/GED [Count of Participants; unit: Participants] | 81 | 73 | 76 | 230
Yearly household income [Count of Participants; unit: Participants]
  Less than $20,000 | 64 | 62 | 63 | 189
  $20,000 to $30,000 | 14 | 19 | 16 | 49
  Greater than $30,000 | 23 | 13 | 10 | 46
  Unknown or Not Reported | 6 | 12 | 8 | 26
Employment [Count of Participants; unit: Participants]
  Not Employed | 55 | 68 | 45 | 168
  Employed Part Time | 21 | 19 | 32 | 72
  Employed Full Time | 30 | 19 | 20 | 69
  Unknown or Not Reported | 1 | 0 | 0 | 1
Married or Living with Partner [Count of Participants; unit: Participants] | 74 | 65 | 64 | 203
Place of Birth [Count of Participants; unit: Participants]
  US 50 States/District of Columbia | 5 | 9 | 6 | 20
  Mexico | 97 | 95 | 89 | 281
  Other | 5 | 2 | 2 | 9
Primary Language is Spanish [Count of Participants; unit: Participants] | 101 | 98 | 90 | 289
Has Some Type of Health Insurance [Count of Participants; unit: Participants] | 53 | 57 | 42 | 152
Health Literacy [Count of Participants; unit: Participants] — Single Item Literacy Scale
  Participants
    Adequate | 56 | 56 | 55 | 167
    Limited | 51 | 50 | 42 | 143
Duration of Diabetes Diagnosis [Mean (Standard Deviation); unit: years] | 10.22 (8.22) | 10.31 (8.25) | 10.59 (8.26) | 10.37 (8.22)
BMI [Mean (Standard Deviation); unit: units kg/m^2] | 31.84 (5.82) | 33.51 (7.35) | 31.37 (6.34) | 32.22 (6.54)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin] | 9.25 (1.64) | 9.31 (1.58) | 9.37 (1.56) | 9.31 (1.59)
Low-density Lipoprotein-cholesterol (LDL-C); [Mean (Standard Deviation); unit: mg/dL] — Population: Sample sizes differ due to missing values.
  mg/dL
    number analyzed (Participants) | 102 | 102 | 95 | 299
    (all) | 93.07 (38.75) | 91.17 (33.88) | 100.32 (41.03) | 94.72 (38.00)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm/Hg] — Population: Sample sizes differ due to missing values.
  mm/Hg
    number analyzed (Participants) | 106 | 104 | 95 | 305
    (all) | 121.36 (17.11) | 122.69 (17.96) | 123.08 (20.10) | 122.35 (18.33)
Patient-Provider Communication [Mean (Standard Deviation); unit: units on a scale] — Patient- provider communication was assessed using the healthcare team subscale of the Chronic Illness Resource Survey (range, 1-5). Higher scores indicate greater perceived support or engagement with the healthcare team (e.g., physicians, nurses, diabetes educators) in managing the chronic illness. Population: Sample sizes differ due to missing values.
  units on a scale
    number analyzed (Participants) | 104 | 102 | 95 | 301
    (all) | 4.06 (1.03) | 3.97 (1.05) | 4.12 (1.02) | 4.05 (1.03)
Patient Blood Glucose Monitoring [Mean (Standard Deviation); unit: days per week] — Population: Sample sizes differ due to missing values.
  days per week
    number analyzed (Participants) | 102 | 95 | 84 | 281
    (all) | 4.11 (1.26) | 4.46 (2.50) | 4.38 (2.83) | 4.31 (2.62)
Participated in Aerobic Exercise [Mean (Standard Deviation); unit: units on a scale] — Aerobic exercise was assessed using the aerobic subscale of the Rapid Assessment of Physical Activity (Seven-point scale, 1-7). Population: Sample sizes differ due to missing values.
  units on a scale
    number analyzed (Participants) | 104 | 98 | 88 | 290
    (all) | 5.01 (1.64) | 5.14 (1.78) | 4.73 (1.67) | 4.97 (1.70)
Participated in Strength Exercise [Count of Participants; unit: Participants] | 25 | 27 | 17 | 69
Participated in Flexibility Exercise [Count of Participants; unit: Participants] | 40 | 54 | 46 | 140
Healthy Eating Behaviors [Mean (Standard Deviation); unit: units on a scale] | 49.63 (6.87) | 50.29 (7.23) | 49.33 (6.88) | 49.76 (6.99)
Diabetes Distress [Mean (Standard Deviation); unit: units on a scale] — Population: Sample sizes differ due to missing values.
  units on a scale
    number analyzed (Participants) | 105 | 101 | 95 | 301
    (all) | 2.39 (1.01) | 2.43 (0.99) | 2.40 (0.97) | 2.41 (0.99)
Adherence to Refills and Medications Scale (ARMS) [Mean (Standard Deviation); unit: units on a scale] — Population: Sample sizes differ due to missing values.
  units on a scale
    number analyzed (Participants) | 104 | 99 | 94 | 297
    (all) | 17.87 (3.99) | 18.28 (5.60) | 18.40 (4.40) | 18.18 (4.70)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin (HbA1c) 6 Months After Enrollment
Description: Glycosylated Hemoglobin (HbA1c) six months after enrollment
Time Frame: 6 months from baseline
Population: Participants that came in for 6-month measures
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Dulce Digital-Me (Medical Assistants): The third of the three arms of the parallel design: The group of participants randomly assigned to this arm of the study receives educational text messages, with patient monitoring and transmission of blood glucose values, plus personalized goal-setting and tailored feedback delivered by Medical Assistants, incorporated into existing primary care team processes.
- Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants): Dulce Digital-Me (Combination of two intervention groups: Automated Delivery and Medical Assistants)
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 77 | 76 | 73 | 149
percentage | 8.17 (1.51) | 7.99 (1.61) | 8.44 (1.48) | 8.21 (1.56)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for age, gender, employment and language; Test type: Superiority; p = 0.95, Regression, Logistic

2. Primary Outcome: Glycosylated Hemoglobin (HbA1c) 12 Months After Enrollment
Description: Glycosylated Hemoglobin (HbA1c) twelve months after enrollment
Time Frame: 12 months from baseline
Population: Participants that came in for 12-month measures
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 67 | 66 | 65 | 131
percentage | 8.29 (1.62) | 8.41 (1.70) | 8.83 (1.83) | 8.62 (1.77)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for age, gender, employment, and language; Test type: Superiority; p = 0.37, Regression, Logistic

3. Primary Outcome: Low-density Lipoprotein-cholesterol (LDL-C); 6 Months After Enrollment
Description: Low-density lipoprotein-cholesterol (LDL-C); six months after enrollment
Time Frame: 6 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 60 | 56 | 58 | 174
mg/dL | 90.27 (33.66) | 88.20 (36.38) | 102.93 (47.96) | 95.69 (43.12)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for age, gender, employment, and language; Test type: Superiority; p = 0.26, Regression, Logistic

4. Primary Outcome: Low-density Lipoprotein-cholesterol (LDL-C); 12 Months After Enrollment
Description: Low-density lipoprotein-cholesterol (LDL-C); twelve months after enrollment
Time Frame: 12 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 41 | 49 | 48 | 138
mg/dL | 97.85 (27.74) | 94.10 (35.18) | 92.04 (43.23) | 93.08 (39.18)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for age, gender, employment, and language; Test type: Superiority; p = 0.90, Regression, Logistic

5. Primary Outcome: Systolic Blood Pressure (SBP); 6 Months From Enrollment
Description: Systolic blood pressure (SBP); six months from enrollment
Time Frame: 6 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 79 | 73 | 72 | 154
mm/Hg | 126.70 (19.52) | 124.84 (18.66) | 124.78 (19.13) | 124.81 (18.83)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for age, gender, employment, and language; Test type: Superiority; p = 0.21, Regression, Logistic

6. Primary Outcome: Systolic Blood Pressure (SBP); 12 Months From Enrollment
Description: Systolic blood pressure (SBP); twelve months from enrollment
Time Frame: 12 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 64 | 67 | 67 | 134
mm/Hg | 125.10 (17.38) | 122.82 (15.29) | 124.13 (19.54) | 123.47 (17.49)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for age, gender, employment, and language; Test type: Superiority; p = 0.30, Regression, Logistic

7. Secondary Outcome: Patient-Provider Communication; 6 Months From Enrollment
Description: Patient-Provider Communication as reported by patient; six months from enrollment The minimum value on the scale is 1 and the maximum value on the scale is 5. A higher score is a better outcome.
Time Frame: 6 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 70 | 64 | 62 | 126
score on a scale | 4.18 (1.05) | 4.04 (1.02) | 4.28 (0.80) | 4.16 (0.92)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.90, Regression, Logistic

8. Secondary Outcome: Patient-Provider Communication; 12 Months From Enrollment
Description: Patient-Provider Communication as reported by patient; twelve months from enrollment The minimum value on the scale is 1 and the maximum value on the scale is 5. A higher score is a better outcome.
Time Frame: 12 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 54 | 60 | 48 | 108
score on a scale | 4.09 (1.03) | 3.99 (1.04) | 4.16 (0.96) | 4.06 (1.00)
Statistical Analysis 1: Comparison: Dulce Digital; Analyses controlled for income; Test type: Superiority; p = 0.72, Regression, Logistic

9. Secondary Outcome: Patient Blood Glucose Monitoring; 6 Months From Enrollment
Description: Patient Blood Glucose Monitoring as reported by patient; six months from enrollment The minimum value on this scale is 1 day per week and the maximum value on this scale is 7 days per week.
  A higher value on this scale is a better outcome.
Time Frame: 6 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 69 | 63 | 61 | 124
days per week | 5.07 (2.29) | 5.62 (1.99) | 5.11 (2.41) | 5.37 (2.21)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.61, Regression, Logistic

10. Secondary Outcome: Patient Blood Glucose Monitoring; 12 Months From Enrollment
Description: Patient Blood Glucose Monitoring as reported by patient; twelve months from enrollment The minimum value on this scale is 1 day per week and the maximum value on this scale is 7 days per week.
  A higher value on this scale is a better outcome.
Time Frame: 12 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 52 | 60 | 48 | 108
days per week | 5.08 (2.19) | 4.77 (2.65) | 5.15 (2.41) | 4.94 (2.54)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.49, Regression, Logistic

11. Secondary Outcome: Participated in Aerobic Exercise; 6 Months From Enrollment
Description: Participated in Aerobic Exercise as reported by patient, six months from enrollment The minimum score is 1 and the maximum score is 7. A higher score is a better outcome.
Time Frame: 6 months from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 68 | 63 | 61 | 124
score on a scale | 5.46 (1.48) | 5.29 (1.50) | 5.49 (1.45) | 5.41 (1.47)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.96, Regression, Logistic

12. Secondary Outcome: Participated in Aerobic Exercise; 12 Months From Enrollment
Description: Participated in Aerobic Exercise as reported by patient, twelve months from enrollment The minimum score is 1 and the maximum score is 7. A higher score is a better outcome.
Time Frame: 12 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 54 | 57 | 47 | 104
score on a scale | 5.11 (1.48) | 5.12 (1.77) | 4.72 (1.94) | 4.94 (1.85)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.64, Regression, Logistic

13. Secondary Outcome: Participated in Strength Exercise; 6 Months From Enrollment
Description: Participated in Strength Exercise as reported by patient; six months from enrollment
Time Frame: 6 months from baseline
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 89 | 85 | 74 | 159
Participants | 20 | 11 | 10 | 21
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Binary logistic analyses were conducted for this outcome. Unstandardized regression coefficients represent logit coefficients; Test type: Superiority; p = 0.87, Regression, Logistic

14. Secondary Outcome: Participated in Strength Exercise; 12 Months From Enrollment
Description: Participated in Strength Exercise as reported by patient; twelve months from enrollment
Time Frame: 12 months from baseline
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 56 | 63 | 51 | 114
Participants | 12 | 9 | 8 | 17
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Binary logistic regression analyses were conducted for this outcome. Unstandardized regression coefficients represent logit coefficients; Test type: Superiority; p = 0.58, Regression, Logistic

15. Secondary Outcome: Participated in Flexibility Exercise; 6 Months From Enrollment
Description: Participated in Flexibility Exercise as reported by patient; six months from enrollment
Time Frame: 6 months from baseline
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 89 | 85 | 74 | 159
Participants | 44 | 39 | 31 | 70
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.25, Regression, Logistic

16. Secondary Outcome: Participated in Flexibility Exercise; 12 Months From Enrollment
Description: Participated in Flexibility Exercise as reported by patient; twelve months from enrollment
Time Frame: 12 months from baseline
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 56 | 63 | 51 | 114
Participants | 29 | 34 | 15 | 49
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.11, Regression, Logistic

17. Secondary Outcome: Healthy Eating Behaviors; 6 Months From Enrollment
Description: Healthy Eating Behaviors as reported by patient; six months from enrollment The minimum score is 20 and the maximum score is 76. The higher score represents a better outcome.
Time Frame: 6 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 89 | 85 | 74 | 159
score on a scale | 50.12 (6.38) | 50.48 (6.96) | 49.41 (6.66) | 49.98 (6.82)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.76, Regression, Logistic

18. Secondary Outcome: Healthy Eating Behaviors; 12 Months From Enrollment
Description: Healthy Eating Behaviors as reported by patient; twelve months from enrollment The minimum score is 20 and the maximum score is 76. The higher score represents a better outcome.
Time Frame: 12 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 56 | 63 | 51 | 114
score on a scale | 51.04 (6.0) | 50.24 (5.81) | 50.67 (6.19) | 50.43 (5.96)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.05, Regression, Logistic

19. Secondary Outcome: Diabetes Distress; 6 Months From Enrollment
Description: Diabetes Distress as reported by patient; six months from enrollment The minimum score is 1 and the maximum score is 6. A higher score represents a worse outcome.
Time Frame: 6 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 70 | 65 | 62 | 127
score on a scale | 2.16 (0.83) | 2.12 (0.93) | 2.16 (0.89) | 2.14 (0.91)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.63, Regression, Logistic

20. Secondary Outcome: Diabetes Distress; 12 Months From Enrollment
Description: Diabetes Distress as reported by patient; twelve months from enrollment The minimum score is 1 and the maximum score is 6. A higher score represents a worse outcome.
Time Frame: 12 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 53 | 60 | 48 | 108
score on a scale | 1.96 (0.75) | 2.23 (0.96) | 2.07 (0.94) | 2.16 (0.95)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses is controlled for income; Test type: Superiority; p = 0.63, Regression, Logistic

21. Secondary Outcome: Adherence to Refills and Medications Scale (ARMS) - Patient-reported Outcome; 6 Months From Enrollment
Description: Adherence to Refills and Medications Scale (ARMS) - Patient-reported Outcome; six months from enrollment The minimum score is 11 and the maximum score is 44. A higher score is a better outcome.
Time Frame: 6 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 70 | 64 | 62 | 126
score on a scale | 17.23 (4.38) | 16.31 (4.04) | 16.12 (3.94) | 16.22 (3.97)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.002, Regression, Logistic

22. Secondary Outcome: Adherence to Refills and Medications Scale (ARMS) - Patient-reported Outcome; 12 Months From Enrollment
Description: Adherence to Refills and Medications Scale (ARMS) - Patient-reported Outcome; twelve months from enrollment The minimum score is 11 and the maximum score is 44. A higher score is a better outcome.
Time Frame: 12 months from baseline
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistants) | Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants)
Number analyzed (Participants) | 53 | 59 | 48 | 107
score on a scale | 16.68 (4.23) | 16.25 (4.26) | 15.85 (3.88) | 16.08 (4.08)
Statistical Analysis 1: Comparison: Dulce Digital vs Dulce Digital-Me (Combined: Automated Delivery and Medical Assistants); Analyses controlled for income; Test type: Superiority; p = 0.008, Regression, Logistic

ADVERSE EVENTS:
Time Frame: From the time of individual patient recruitment at baseline through the end of month 12.
Description: The one all-cause mortality event was discovered when attempting to reach a participant to complete the 12-month measures.
Arm/Group | Dulce Digital | Dulce Digital-Me (Automated Delivery) | Dulce Digital-Me (Medical Assistant)
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/106 | 1/97
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/106 | 0/97
Other Adverse Events (participants affected / at risk) | 0/107 | 0/106 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT03130699/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03130699/ICF_001.pdf